CLINICAL TRIAL: NCT07156669
Title: Safety and Performance of the Novalung Ultimate Kit and Xenios 2.0 During Stationary Use in Hospital and Ground-based Transport of Patients on Extracorporeal Life Support (ECLS)
Acronym: Transport+
Status: Not yet recruiting | Type: Observational
Sponsor: Xenios AG (Industry)
Collaborators: Alcedis GmbH (Industry)
Responsible Party: Sponsor
Organization: Fresenius Medical Care Deutschland GmbH (Industry)
Other Study IDs: HL-ECMO-01-INT
Record Dates: First submitted 2025-06-05; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Cardio-Respiratory Failure; Extracorporeal Membrane Oxygenation Complication; Acute Lung Injury
Keywords: Extracorporeal Life Support; Extracorporeal Membrane Oxygenation
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Extracorporeal Life Support (ECLS): Patients who receive ECLS treatment and require a ground-based inter- hospital patient transport and/ or stationary treatment on ECMO
  Interventions: Device: Novalung ultimate kit, Xenios 2.0, and MultiSupport Ground (MSG)

INTERVENTIONS:
Device: Novalung ultimate kit, Xenios 2.0, and MultiSupport Ground (MSG) — Patients will receive ECLS treatment using the Novalung ultimate kit, Xenios 2.0, and MultiSupport Ground (MSG) during ground-based inter-hospital patient transport and/ or stationary treatment according to their intended use and local standards/ requirements.

SUMMARY:
This prospective observational study will evaluate the safety and performance of the Novalung ultimate kit in combination with the Xenios 2.0 and the MultiSupport Ground during stationary use in hospital and ground-based transport of patients treated on extracorporeal membrane oxygenation (ECMO). The primary objective is to assess whether the use of the medical devices improves and maintains the gas exchange (blood oxygenation) in these patients. Medical Devices will be used according to their intended purpose and local standards/ requirements.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients receiving an ECMO treatment with the Novalung ultimate kit in combination with the Xenios 2.0 (and the MultiSupport Ground during inter- and intra-hospital transport, if applicable) according to the intended use
* Informed consent signed and dated by the attending physician; and

  1. If patient is able to give consent: by the study patient
  2. If patient is unable to give consent: by the legal representative or
  3. If an emergency situation is determined: by a consultant physician

Exclusion Criteria:

* Participation in any interventional clinical study that could impact the results of this prospective, observational PMCF study
* Previous participation in the same study
* ECMO cannulation outside the referring or trial site hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe acute respiratory and/or cardiopulmonary failure treated on ECMO.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Arterial oxygen saturation (SaO2) [%] | Baseline and during the ECMO treatment every 24 hours until a maximum of 29 days
  Longitudinal assessments of continuous outcomes will be analyzed by treatment day using mixed models for repeated measures (MMRM), with ECMO mode as a fixed factor (except for analyses performed within the subsets defined by ECMO mode) and the baseline value of the primary endpoint as a covariate.
  Within-subject differences between baseline and subsequent visits will be tested using contrasts. The comparison between baseline and the first day on ECMO (initial effect) is considered as the primary outcome.

SECONDARY OUTCOMES:
Performance objective Cardiacirculation | Baseline and during the ECMO treatment every 24 hours until a maximum of 29 days
  Improvement and maintenance of patients' cardiocirculation in patients transported and treated stationary on ECMO
Performance objective Maintenance of blood flow | Baseline and during the ECMO treatment every 24 hours until a maximum of 29 days
  Evaluation of Xenios 2.0 performance during transport and stationary use: Maintenance of blood flow (L/min)
Performance objective Pump speed | Baseline and during the ECMO treatment every 24 hours until a maximum of 29 days
  Evaluation of Xenios 2.0 performance during transport and stationary use: Pump speed (rpm)
Performance objective Circuit pressures | Baseline and during the ECMO treatment every 24 hours until a maximum of 29 days
  Evaluation of Xenios 2.0 performance during transport and stationary use: Circuit pressures (mmHg)
Safety objectives | Baseline and during the ECMO treatment every 24 hours until a maximum of 29 days
  Assessment of the safety of the use of the Xenios System for ground-based transport and stationary use of patients on ECMO.
  Complications will be grouped in device-, transport-, cannula-, and patient-related complications and presented as relative and absolute frequencies.

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Groesdonk, Prof. Dr. med., Principal Investigator — HELIOS Hospital, Erfurt, Germany

IPD SHARING:
Plan to Share IPD: Undecided